CLINICAL TRIAL: NCT06623604
Title: The Effect of the Physical Activity Program Developed According to the Precede-Proceed Model on the Physical Activity Level and Physical Activity Behavior of Elementary School Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Muğla Sıtkı Koçman University (Other)
Collaborators: Ege University (Other)
Responsible Party: Principal Investigator, Recep Kara, Research Assistant PHD, Muğla Sıtkı Koçman University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: MuglaSKURK
Record Dates: First submitted 2024-09-19; First posted 2024-10-02 (Actual); Last update posted 2024-10-02 (Actual); Status verified 2024-09

CONDITIONS: Physical Activity; Physical Activity Levels; Physical Activity Behavior
Keywords: Precede-proceed model; school nursing; physical activity; child
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Intervention Model Description: In consultation with school administrators and classroom teachers, a physical activity program was implemented so that students&amp;amp;amp;amp;amp;amp;#39; classes would not be disrupted. Exercises in the program include light and moderate movements that may be performed by a healthy student between the ages of 9 and 11. Sport physicians have advised that there is no need for any health screening, as children&amp;amp;amp;amp;amp;amp;#39;s hearts, pulses, and muscles are not affected by light and moderate exercises. The exercises were carried out three days a week for 30 minutes in the school garden and gym by the same researcher, and the education was carried out in the classrooms one day a week. The researcher performing the exercises received education in an earlier study that included physical exercises and yoga movements. During the program, students did a total of 180 hours of physical activity.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Physical Activity Program (Experimental): The physical activity program consists of two parts: exercise and education. Exercises in the program include light and moderate movements that may be performed by a healthy student between the ages of 9 and 11. The exercises were carried out three days a week for 30 minutes in the school garden and gym by the same researcher, and the education was carried out in the classrooms one day a week. During the program, students did a total of 180 hours of physical activity. In addition, the students' teachers also participated in the program and did exercises with their students. Throughout the program, exercises included 'belly and abdominal movement sets' in the first four weeks, 'leg and hip movement sets' in the following four weeks, and 'arms, shoulder, and chest movement sets' in the final four weeks, as well as yoga movements.
  Interventions: Behavioral: Experimental: Physical activity program
- Control Group (No Intervention): Measurements and questionnaires were applied to the control group.

INTERVENTIONS:
Behavioral: Experimental: Physical activity program — In consultation with school administrators and classroom teachers, a physical activity program was implemented so that students' classes would not be disrupted.
  The exercises were carried out three days a week for 30 minutes in the school garden and gym by the same researcher, and the education was carried out in the classrooms one day a week.
  During the program, students did a total of 180 hours of physical activity.
  Arms: Physical Activity Program

SUMMARY:
The present study aims to investigate the effect of the physical activity program developed according to the Precede-Proceed Model on children's physical activity level and physical activity self-efficacy, attitude, enjoyment level, and exercise change behaviors. This study was conducted in an experimental design with a pretest-posttest control group. Considering the possibility of data loss during the research, 178 students between the ages of 9 and 11 were included in the study, 89 in the intervention group and 89 in the control group. The exercises were carried out three days a week for 30 minutes in the school garden and gym, and the training was carried out in the classrooms one day a week.

ELIGIBILITY:
Inclusion Criteria:

* Enrolled in the fourth grade at the designated schools
* Could read and write
* Families agreed to participate and gave their consent

Exclusion Criteria:

* Have chronic and metabolic diseases or disabilities

Ages: 9 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 89 (Actual)
Dates: Start 2021-10-24 (Actual); Primary Completion 2022-03-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Physical Activity Self-Efficacy Scale (PASS) | 0-6 months
  Physical Activity Self-Efficacy Scale (PASS) was used to measure the physical self-efficacy of children.
Attitude toward Physical Activity Scale (APAS) | 0-6 months
  Attitude toward Physical Activity Scale (APAS) was used to measure the physical activity attitude of children.
Physical Activity Levels | 0-6 months
  The Physical Activity Questionnaire for Older Children (PAQ-C) was used to measure the physical activity level of children.

CONTACTS AND LOCATIONS:
Overall Officials: Recep KARA, Ph.D, Principal Investigator — Muğla Sıtkı Koçman University
Locations (1):
- Muğla Sıtkı Koçman University, Fethiye, Muğla, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No